CLINICAL TRIAL: NCT06520982
Title: Early Neurovascular Adaptations in Aging Women
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American Heart Association (AHA) (Unknown)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Associate Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2109189
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Women; Sympathetic Nervous System; Aging; Blood Flow
MeSH Terms: interventions — Norepinephrine; Isoproterenol; Acetylcholine; Nitroprusside; Estrogens

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Women (Other): Women will be 18-70 years of age
  Interventions: Drug: Norepinephrine; Drug: Isoproterenol; Drug: Acetylcholine; Drug: Nitroprusside; Drug: Estrogen

INTERVENTIONS:
Drug: Norepinephrine — Infused intra-arterially in a dose-response fashion
Drug: Isoproterenol — Infused intra-arterially in a dose-response fashion
Drug: Acetylcholine — Infused intra-arterially in a dose-response fashion
Drug: Nitroprusside — Infused intra-arterially in a dose-response fashion
Drug: Estrogen — Infused intra-arterially

SUMMARY:
Our goal is to enhance our understanding of early vascular adaptations in aging women with an emphasis on the sympathetic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth (AFAB)
* 18-70 years of age

Exclusion Criteria:

* Assigned male at birth (AMAB)
* Pregnancy, breastfeeding
* Body mass index ≥30 kg/m2
* Taking medications known to affect metabolic, autonomic, and/or respiratory function
* Oral hormonal contraception in last 6 month
* History of hormone replacement therapy
* History of hyster- or oophor-ectomy
* Current smoking/Nicotine use
* Increased risk of bleeding, pro-coagulant disorders, clotting disorders, anticoagulation therapy
* Chronic disease
* Blood pressure ≥140/90 mmHg
* Communication barriers

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Magnitude of forearm blood flow | Change from baseline during infusion

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No